CLINICAL TRIAL: NCT02763410
Title: Impact of the Composition of the Packed Red Blood Cell Supernatant on Renal Dysfunction and Post-transfusion Immunomodulation
Brief Title: Impact of the Composition of Packed Red Blood Cell Supernatant on Renal Dysfunction and Posttransfusion Immunomodulation
Acronym: TRANSNEPHRON
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0420
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples and PRBC tubing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control group: Patients who received between 1 and 5 PRBCs between incision and the 6th hour post-surgery, with no renal failure at the 48th hour after surgery, based on the RIFLE classification, and regardless of the transfusion received after the H6 assessment.
  Interventions: Other: PRBC transfusion
- Renal failure group: Patients who received between 1 and 5 PRBCs between incision and the 6th hour post-surgery and who developed renal failure before H48 with no new transfusion prior to diagnosis of kidney failure.
  Interventions: Other: PRBC transfusion

INTERVENTIONS:
Other: PRBC transfusion

SUMMARY:
Safety during transfusions is a major issue in medical economics. Despite drastic quality control measures, transfusion is still a source of short, mid and long-term morbi-mortality. This can be explained to some extent by changes in the composition of the packed red blood cell (PRBC) supernatant during storage essentially with the appearance of immunologically active compounds possibly involved in organ dysfunction on the one hand and post-transfusion immunomodulation on the other hand. These phenomena impact upon outcomes for cardiac surgery patients.

In terms of organ dysfunction, kidney failure due to acute tubular necrosis and pulmonary failure are the 2 main issues. Following cardiac surgery, 11% of patients will present with transient renal dysfunction characterised by a 25% increase in serum creatinine levels and 3.5% require dialysis. The intensity of acute renal failure (ARF) is correlated to resuscitation : a 20% increase in serum creatinine levels 2 to 3 days after surgery significantly raises morbidity rates and a 50% increase raises the mortality rate to 10%.

The precise mechanisms governing post-transfusion immunomodulation have not yet to be defined. The appearance of soluble type I Human leukocytes Antigen (HLA) molecules (sHLA-I), the FAS ligand (FAS-L) or cluster designation 40 (CD40-L) in the supernatant of PRBCs along the storage of blood products may be involved in such phenomena. These molecules are capable of activating or triggering the death of innate or adaptive immunity cells, especially the Natural Killer (NK) cells.

Consequently the investigators propose to focus specifically on the detailed composition of transfused PRBC supernatants in order to identify the candidate molecules responsible for organ dysfunction or post-transfusion immunoparalysis. The investigators will combine a clinical approach based on the transcriptional analysis of renal tubular cells in transfused patients and an ex-vivo approach investigating the effect of the supernatant on immune cells and the Natural Killer cells of healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Non-emergency cardiac surgery under extracorporeal circulation (CEC) with cardioplegia:

And no indication of pre-surgical PRBC transfusion (priming excluded), And no indication of transfusion with fresh frozen plasma or pre-surgical platelet concentrate

Exclusion Criteria:

* Heart and/or lung transplant surgery;
* Emergency surgery to be performed within 24 hours;
* Patient <18 years old;
* Pregnant woman
* Protected adult
* Adult incapable of expressing his/her non-opposition
* Opposition expressed by the patient on recording his/her data;
* No French social security;
* Patient who underwent a transfusion in the 3 months prior to surgery;
* Surgery due to endocarditis or suspected endocarditis;
* Myocardial infarction < 15 days;
* Patient receiving inotropic or vasopressor prior to surgery;
* Patient receiving immunosuppressant treatment;
* Patient receiving corticosteroids for 21 days or more;
* Seropositive patient known to be suffering from HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Currently taking antibiotics (except permitted peri-surgical antibiotic prophylaxis );
* History of advancing cancer;
* Clearance < 40 ml/min/m2 according to the Modification of Diet in Renal Disease (MDRD) during the pre-surgical assessment;
* Positive irregular antibody test warranting a cross-match prior to transfusion.
* Patients with indwelling urinary catheter preoperatively
* preoperative positive urine culture
* Urinary tract infection <21 days before surgery
* Background gesture on the upper or lower urinary tract

Exclusion criteria analysis

* In the renal insufficient group: Patient transfused plasma (s) Fresh Frozen (s) (PFCs) or concentrate (s) platelet (s) (CP) after the balance sheet T6 (6 hours after arrival in the ICU) and before the diagnosis of ARF,
* strict anuric patient not to achieve a 50 ml urine sample at least
* Reversal surgery requiring CEC before the 48th hour
* Surgical Complication could explain the acute renal failure (IRA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients:
  The investigators selected cardiac surgery patients for the transfusion frequency and significant post-surgical renal morbidity.
  Study centre:
  The study will take place at the CHU Nantes (University Hospital Centre) where over 1500 extracorporeal circulation procedures are performed annually.
  Number of patients required: 200 patients:
  100 transfusion patients who have developed renal failure; 100 transfusion patients who have not developed renal failure;
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
link between the composition of the PRBC supernatant and the onset of renal failure | 48 hours following surgery

SECONDARY OUTCOMES:
Respiratory dysfunction in the ICU defined by a blood pressure of oxygen (PaO2)/inspired oxygen fraction (FiO2) ratio < 300 on at least one occasion | within 28 days
Number of dialysis days | within 28 days
Duration of stay | within 28 days
Ventilation period (in hours); | within 28 days
ICU-acquired infection | within 28 days
Status at discharge from ICU: Dead/alive | day 28
Study of transfusion-related accidents recorded in ICU | within 28 days
Hospital admission, regardless of cause | 1 year
Hospital admission due to infection | 1 year
Diagnosis of cancer | 1 year
Clinical course of pre-existing cancer | 1 year
Survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France